CLINICAL TRIAL: NCT00502632
Title: Multicentre Randomized Double-Blinded Trial of Intrapleural Dornase Alfa and Urokinase vs Urokinase Alone for Complicated Parapneumonic Effusions in Children
Brief Title: Dornase Alfa and Urokinase for Kids With Pleural Empyema
Acronym: DUKE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr PierGiorgio Gamba, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1372P
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Pleural Empyema
Keywords: Pleural empyema; Pleural effusion; Dornase alfa; Urokinase; Children
MeSH Terms: conditions — Empyema, Pleural; Pleural Effusion | interventions — Urokinase-Type Plasminogen Activator; dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intrapleural administration of:
  * Urokinase 40,000 in 40ml normal saline, twice daily for 4 days
  * Dornase alfa 2,500 IU in 25ml normal saline, twice daily for 4 days
  Interventions: Drug: Urokinase and Dornase alfa
- 2 (Placebo Comparator): Intrapleural administration of:
  * Urokinase 40,000 in 40ml normal saline, twice daily for 4 days
  * 25ml normal saline, twice daily for 4 days
  Interventions: Drug: Urokinase

INTERVENTIONS:
Drug: Urokinase and Dornase alfa — Intrapleural administration of:
  * Urokinase 40,000 in 40ml normal saline, twice daily for 4 days
  * Dornase alfa 2,500 IU in 25ml normal saline, twice daily for 4 days
  Arms: 1
Drug: Urokinase — Intrapleural administration of:
  * Urokinase 40,000 in 40ml normal saline, twice daily for 4 days
  * 25ml normal saline, twice daily for 4 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether intrapleural treatment with Dornase alfa plus Urokinase improves clinical outcome compared to Urokinase alone in children with complicated parapneumonic effusions

ELIGIBILITY:
Inclusion Criteria:

* Age > 1 year and < 16 years
* Respiratory infection (pneumonia or lung abscess)
* Effusion occupying at least 1/3 of hemithorax on chest X-ray
* Complicated effusion (presence of at least one of the following):

  * Hyperechoic pleural fluid on chest US scan
  * Loculated collection on chest US or CT scan
  * Purulent pleural fluid
  * Positive culture or Gram stain on pleural fluid

Exclusion Criteria:

* Non parapneumonic effusion
* Immunodeficiency
* Neurological impairment
* Suspected or proven allergy to Urokinase or Dornase alfa
* Suspected or documented bronchopleural fistula
* Impaired coagulation (INR>2), haemorrhage, high risk for bleeding
* Thoracic surgical procedure (e.g. thoracoscopy, mini-thoracotomy) already performed
* Chest drain inserted since 6 or more days

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2007-10; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay | From beginning of intrapleural treatment
Need for additional surgical procedures | 3 months

SECONDARY OUTCOMES:
Duration of suction applied to chest drain | From beginning of intrapleural treatment
Duration of fever | From beginning of intrapleural treatment
Duration of intravenous antibiotic treatment | From beginning of intrapleural treatment

CONTACTS AND LOCATIONS:
Overall Officials: PierGiorgio Gamba, MD, Study Chair — Azienda Ospedaliera di Padova; Giorgio Stefanutti, MD, Principal Investigator — Women's and Children's Hospital, Adelaide, SA
Locations (3):
- Italy (3):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Bambino Gesu', Roma